CLINICAL TRIAL: NCT05631574
Title: A Phase 1/1b Dose Finding Study of BMF-219, an Oral Covalent Menin Inhibitor, in Adult Patients With Unresectable, Locally Advanced, or Metastatic Non-small Cell Lung Cancer (NSCLC), Pancreatic Cancer (PDAC), and Colorectal Cancer (CRC)
Brief Title: Study of Covalent Menin Inhibitor BMF-219 in Adult Patients With KRAS Driven Non-Small Cell Lung Cancer, Pancreatic Cancer, and Colorectal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Biomea Fusion, Inc., is no longer pursuing oncology indications for BMF-219. No safety concerns or efficacy observations led to this study closure.
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: COVALENT-102
Record Dates: First submitted 2022-11-04; First posted 2022-11-30 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Non Small Cell Lung Cancer; Pancreatic Cancer; Colorectal Cancer; NSCLC; PDAC; CRC; Relapsed Cancer; Refractory Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer; Stage III Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Stage III Colorectal Cancer; Stage IV Colorectal Cancer; Stage III NSCLC; Stage IV NSCLC; KRAS Mutation-Related Tumors
Keywords: Oral Covalent Menin Inhibitor; Relapsed; Refractory; Irreversible Menin Inhibitor; Menin Inhibitor; Unresectable; Locally Advanced; Metastatic; Menin; Menin Therapy; KRAS; KRAS Mutated
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Colorectal Neoplasms; Recurrence; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This study is an ascending multiple dose clinical trial followed by cohort expansion. The dose escalation part is primarily intended to identify the optimal biologic dose (OBD)(s) of BMF-219 and to obtain initial safety and tolerability information regarding the compound when administered orally to subjects with KRAS mutated unresectable, locally advanced, or metastatic NSCLC, PDAC and CRC. This study will also evaluate the PK/PD profiles of multiple dose administration of BMF-219. Following completion of the dose escalation, cohort and arm-specific expansion cohorts will commence in order to further confirm the safety and tolerability of BMF-219 dosed at or near the OBD.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation Phase (Experimental): Dose Escalation Phase will group all disease indications (NSCLC, PDAC, and CRC) together to assess the safety of each dose level.
  Participants will receive escalating dose BMF-219 orally once per day or twice per day to identify the OBD/RP2D (Optimal Biologic Dose/Recommended Ph2 Dose).
  Interventions: Drug: BMF-219
- Expansion Phase (Experimental): Dose Expansion Phase will enroll additional subjects independently in each disease indication:
  Cohort 1: Participants with NSCLC
  Cohort 2: Participants with PDAC
  Cohort 3: Patients with CRC
  Cohorts 1, 2, and 3 will receive BMF-219 at the OBD/ RP2D to further assess the safety and efficacy of the investigational drug.
  Interventions: Drug: BMF-219

INTERVENTIONS:
Drug: BMF-219 — BMF-219 is an orally bioavailable, covalent small-molecule menin inhibitor.

SUMMARY:
A Phase 1/1b dose finding study to determine the OBD(s) and RP2D(s) of BMF-219, a covalent menin inhibitor small molecule, in subjects with KRAS mutated unresectable, locally advanced, or metastatic NSCLC (Cohort 1), PDAC (Cohort 2), and CRC (Cohort 3).

DETAILED DESCRIPTION:
This is a dose finding study to determine the safety and tolerability, pharmacokinetics and pharmacodynamics, and clinical activity of escalating doses of BMF-219 administered orally (PO) either once daily (QD) or twice daily (BID) in 28-day cycles. After observing acceptable safety performance in these dosing regimens, additional subjects will be enrolled to assess efficacy in the determination of the OBD for use as a RP2D.

ELIGIBILITY:
Inclusion Criteria

1. Adults with a confirmed diagnosis of unresectable, locally advanced and/or metastatic Stage IIIB/IV NSCLC, Stage III/IV PDAC and/or Stage III/IV CRC with no curative-intent treatment options and documented activating KRAS mutation (without known additional actionable driver mutations such as EGFR, ALK or ROS1)
2. Documented progression and measurable disease after ≥ 1 prior line of systemic therapy (≥ 2 and

   ≤ 4 prior lines for NSCLC) with adequate washout period and resolution of treatment-related toxicities to ≤ Grade 2
3. ECOG PS of 0-2 (0-1 for PDAC) and a life expectancy > 3 months in the opinion of the Investigator
4. Adequate hematological, liver, and renal function
5. Men and women of childbearing potential must use adequate birth control measures for the duration of the trial and at least 90 days after discontinuing study treatment

Exclusion Criteria

1. Symptomatic and/or untreated CNS or brain metastasis, pre-existing ILD or pericardial/pleural effusion of ≥ grade 2 or requiring chronic oxygen therapy for COPD or pleural effusions
2. Serious concomitant disorder including infection
3. Known positive test for HIV, HCV, HBV surface antigen
4. Concurrent malignancy in the previous 2 years
5. Prior menin inhibitor therapy
6. Requiring treatment with a strong or moderate CYP3A inhibitor/inducer
7. Significant cardiovascular disease or QTcF or QTcB prolongation.
8. Major surgery within 4 weeks prior to first dose
9. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
To determine the OBDs/RP2Ds of BMF-219 monotherapy in subjects with KRAS-driven unresectable, locally advanced, or metastatic NSCLC, PDAC and CRC. | 30 months
  OBD/RP2D as determined by the number of subjects receiving BMF-219 monotherapy who experience Dose-Limiting Toxicities (DLTs) within each dose level. A DLT is defined as any clinically significant Adverse Event within 28 days of starting BMF-219 treatment and considered to be related to the IMP. Adverse Events will be assessed per CTCAE v5.0.
To determine the OBDs/RP2Ds of BMF-219 monotherapy in subjects with KRAS-driven unresectable, locally advanced, or metastatic NSCLC, PDAC and CRC. | 30 months
  OBD/RP2D as measured by objective response rate (ORR). ORR will be assessed using RECIST 1.1 per investigator assessment.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of BMF-219 monotherapy. | 46 months
  Safety and tolerability will be determined using treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) as outcomes.
To evaluate the pharmacokinetics of BMF-219. | 46 months
  Pharmacokinetics will be determined using maximum observed plasma concentration (Cmax ).
To evaluate the pharmacokinetics of BMF-219. | 46 months
  Pharmacokinetics will be determined time to maximum plasma concentration (tmax).
To evaluate the pharmacokinetics of BMF-219. | 46 months
  Pharmacokinetics will be determined using the AUC from time 0 to last quantifiable concentration (AUClast ).
To evaluate the efficacy of BMF-219 monotherapy in subjects with unresectable, locally advanced, or metastatic NSCLC, PDAC and CRC. | 46 months
  Efficacy will be determined using duration of response (DOR), defined by the duration of time from the date of initial response of PR or better to the date of disease progression or death due to any cause, whichever occurs first. DOR will be assessed using RECIST 1.1 per investigator assessment.
To evaluate the efficacy of BMF-219 monotherapy in subjects with unresectable, locally advanced, or metastatic NSCLC, PDAC and CRC. | 46 months
  Efficacy determined by disease control rate (DCR), defined as the proportion of response-evaluable subjects who maintain disease control (Complete Response, Partial Response or SD as per RECIST 1.1) from first dose through Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Morris, MD, Study Director — Biomea Fusion Inc.
Locations (23):
- United States (19):
  - Cancer Treatment Centers of America - Phoenix, Goodyear, Arizona
  - California Cancer Associates for Research and Excellence (cCARE), Encinitas, California
  - University of California, San Diego, La Jolla, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Cancer Treatment Centers of America - Atlanta, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern Univeristy, Chicago, Illinois
  - Cancer Treatment Centers of America - Chicago, Zion, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul